CLINICAL TRIAL: NCT04568590
Title: Cohort Study to Determine the Effect of an Educational Intervention Focusing on Herd Immunity to Enhance Vaccination Uptake Rates
Brief Title: Promoting Altruism to Enhance Vaccine Acceptance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00068446
Record Dates: First submitted 2020-09-17; First posted 2020-09-29 (Actual); Results first posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2022-07

CONDITIONS: Vaccine Refusal
Keywords: altruism; vaccine acceptance; flu vaccine
MeSH Terms: conditions — Vaccination Refusal; Altruism; Influenza, Human | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vaccine Hesitant (Experimental): Subjects who consent to this study and deemed vaccine hesitant, they will receive an educational intervention.
  Interventions: Behavioral: educational intervention

INTERVENTIONS:
Behavioral: educational intervention — If the guardian screens positive for vaccine hesitancy (i.e., vaccine hesitancy score average > 3), they will be given the informational handout along with a brief script.

SUMMARY:
Subjects enrolled in this study are eligible for the seasonal influenza vaccine. The purpose of this research study is to figure out if increasing individuals' awareness of the benefits of herd immunity, specifically to the local pediatric oncology community, can improve vaccination uptake rates.

DETAILED DESCRIPTION:
The purpose of this study is to identify associations with influenza vaccine hesitancy, including parental demographics and altruism score, in families with healthy children attending two pediatric practices.

Also, in the cohort of families with baseline vaccine hesitancy, to assess the effectiveness of a pilot educational intervention focusing on the development of herd immunity for pediatric oncology patients by measuring:

1. The change in vaccine hesitancy scores pre- and post-intervention.
2. The rate of influenza vaccine uptake compared to historic controls from previous influenza seasons.

Another aim is to explore the relationship between baseline influenza vaccine hesitancy rates and baseline altruism scores. Effectiveness of this intervention is dependent on parental altruism levels; therefore, the study team also seeks to determine if there is an association between parental altruism and vaccine hesitancy for their children.

This is a single-arm prospective cohort study. The study will enroll legal guardians of children who are influenza vaccine-eligible to measure their vaccine hesitancy scores, altruism scores, and the impact of an educational intervention focused on herd immunity on the guardians' vaccine hesitancy score.

ELIGIBILITY:
Inclusion Criteria:

* All legal guardians of children aged 6 months and up who are influenza vaccine-eligible and present to the pediatric clinic.

Exclusion Criteria:

* Legal guardians of children who are not influenza vaccine-eligible including children less than 6 months of age, children on immunosuppressive medications, and children with underlying medical conditions resulting in an immunocompromised state.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 510 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2021-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Halvorson, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Univesity Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification, will be available. The Study Protocol, Statistical Analysis Plan, and Informed Consent Form will also be available. All data will be available beginning 9 months and ending 36 months following article publication. The study team intends to share with researchers who provide a methodologically sound proposal to achieve aims in the approved proposal. Proposals may be submitted up to 36 months following article publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: All data will be available beginning 9 months and ending 36 months following article publication.
Access Criteria: Please contact PI to request access to data beginning 9 months and ending 36 months after article publication.

REFERENCES:
- [Derived] Marlowe E, Pranikoff S, Borsheim B, Salafian K, Halvorson EE, Kram DE. Pilot study to determine effect of an altruism intervention focusing on herd immunity to enhance influenza vaccination rates. Vaccine. 2022 Nov 2;40(46):6625-6630. doi: 10.1016/j.vaccine.2022.09.074. Epub 2022 Oct 6. PMID 36210252

RESULTS

PARTICIPANT FLOW:
Groups:
- Vaccine Hesitant: Only the Subjects who consent to this study and deemed vaccine hesitant, they will receive an educational intervention.
  educational intervention: If the guardian screens positive for vaccine hesitancy (i.e., vaccine hesitancy score average > 3), they will be given the informational handout along with a brief script.
Period: Overall Study
Arm/Group | Vaccine Hesitant
Started | 510
Completed | 73
Not Completed | 437
Not completed — Subjects were not Vaccine-hesitant | 437

BASELINE CHARACTERISTICS:
Arm/Group | Vaccine Hesitant
Number analyzed (Participants) | 73
Age, Continuous [Mean (Standard Deviation); unit: years] — Age not collected Population: Age not collected
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender data not collected
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 23
  White | 41
  More than one race | 0
  Unknown or Not Reported | 7
Region of Enrollment [Number; unit: participants]
  United States | 73

OUTCOME MEASURES:

1. Primary Outcome: Change in Vaccine Hesitancy Scores Pre- and Post-Intervention.
Description: 8-item Vaccine Hesitancy Scale. Subjects identified as vaccine-hesitant based on a Vaccine Hesitancy Score >/= 3. Score range is 1-5 and > or = 3 is considered vaccine hesitant.
Time Frame: Baseline (Pre-intervention) and Post-Intervention, up to 4 hours
Population: Population who scored as vaccine hesitant initially who completed both the pre-intervention (N=73) and post-intervention (N=68) aVHS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vaccine Hesitant
Number analyzed (Participants) | 68
units on a scale | -0.4 (0.63)

2. Primary Outcome: Pre-Intervention Vaccine Hesitancy Score
Description: as for outcome 1
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vaccine Hesitant
Number analyzed (Participants) | 73
units on a scale | 3.81 (0.61)

3. Primary Outcome: Post-Intervention Vaccine Hesitancy Score
Description: as for outcome 1
Time Frame: Post-Intervention up to 4 Hours
Population: Of our vaccine-hesitant cohort (N=73), only 68 completed the post-intervention aVHS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vaccine Hesitant
Number analyzed (Participants) | 68
units on a scale | 3.42 (0.87)

4. Secondary Outcome: Rate of Influenza Vaccine Uptake
Description: The subject's child's electronic health record will be accessed to document whether that patient received the seasonal influenza vaccine during the baseline visit.
Time Frame: baseline
Population: We examined this outcome for subjects who completed both the pre-intervention (N=73) and post-intervention (N=68) aVHS
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine Hesitant
Number analyzed (Participants) | 68
Participants | 8

5. Secondary Outcome: Pre-Intervention Altruism Scale
Description: Scale ranges from 20-100 with a higher score denoting higher altruism.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vaccine Hesitant
Number analyzed (Participants) | 68
score on a scale | 60.4 (13.3)

6. Other Pre Specified Outcome: Complex Interaction Interviews
Description: Motivational interviews will be conducted with 20 vaccine-hesitant participants, and with four study volunteers. Each motivational interview will be conducted by the same person. Data from these interviews will be entered directly into a Research Electronic Data Capture database and analyzed using Statistical Analysis Software (SAS v9.4).
Time Frame: Month 9
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to one year
Description: No adverse events were anticipated in this trial in which the only intervention was the provision of vaccine information.
Arm/Group | Vaccine Hesitant
All-Cause Mortality (participants affected / at risk) | 0/510
Serious Adverse Events (participants affected / at risk) | 0/510
Other Adverse Events (participants affected / at risk) | 0/510

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-27): https://cdn.clinicaltrials.gov/large-docs/90/NCT04568590/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-13): https://cdn.clinicaltrials.gov/large-docs/90/NCT04568590/ICF_001.pdf